CLINICAL TRIAL: NCT04435197
Title: Multicenter Preoperative Anti-PD-1 Antibody Combined With Chemoradiotherapy for Locally Advanced Squamous Cell Carcinoma of Esophageus
Brief Title: Pre-Operative Pembrolizumab + Chemoradiation in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma
Acronym: PALACE-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Fujian Medical University Union Hospital (Other); Zhejiang University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Chair of thoracic department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-010
Record Dates: First submitted 2020-06-14; First posted 2020-06-17 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Immunotherapy; Pathologic complete response; preoperative pembrolizumab with concurrent chemoradiotherapy; Disease-free Survival; Median overall survival
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Pathologic Complete Response | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Participants will receive carboplatin (AUC=2) IV and paclitaxel (50mg/m²) IV on day 1,8,15,22,29. And radiotherapy will start on day 1 of chemotherapy. A total of 41.4 Gy, 23 fractions of 1.8 Gy, 5 fractions a week. Participants will also receive pembrolizumab (2mg/kg) IV on days 1 and 22. Surgery will be performed within 4-6 weeks after completion of preoperative therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Arm 1:
  A: Pembrolizumab 200mg(100mg if weight less than 50kg) IV on days 1 and 22 B: Carboplatin (AUC=2) IV and paclitaxel (50mg/m²) IV on day 1,8,15,22,29. C: Radiotherapy will start on day 1 of chemotherapy. A total of 41.4 Gy, 23 fractions of 1.8 Gy, 5 fractions a week.
  D: Ivor-Lewis or McKeown esophagectomy
  The participants will receive preoperative A+B+C. 4-6 weeks after completion of preoperative therapy ，D will be performed if there is no contraindication.
  Interventions: Drug: Pembrolizumab Injection

INTERVENTIONS:
Drug: Pembrolizumab Injection — Pre-operative Pembrolizumab+chemoradiotherapy
  Other Names: Keytruda

SUMMARY:
To investigate the safety and activity of preoperative pembrolizumab combined with chemoradiotherapy for resectable esophageal squamous cell carcinoma (ESCC) ,20 patients enrolled in Phase Ib PALACE-1(NCT03792347).The results showed that preoperative pembrolizumab with concurrent chemoradiotherapy was safe, did not delay surgery and induced a pCR in 55.6% of resected tumors. In this multicentre prospective study(PALACE-2),the investigators will evaluate the efficacy of preoperative pembrolizumab with concurrent chemoradiotherapy in patients with locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
For locally advanced esophageal squamous cell carcinoma (ESCC), neoadjuvant chemoradiotherapy followed by surgery has been recommended as the optimal therapeutic strategy.Patients who achieved pathologic complete response(pCR) after receiving neoadjuvant therapy were more likely to have better survival. And the pCR rates was 43.2% reported in NEOCRTEC5010 trial, 49% with ESCC in the CROSS trial and 33.3% in FFCD 990130.

In Phase Ib PALACE-1(NCT03792347), the investigators firstly present that preoperative pembrolizumab combined with chemoradiotherapy followed by surgery is safe.All 20 patients have received PPCT successfully, except 1 patient who missed the last dose of chemotherapy due to leukopenia. Grade 3 and higher adverse events (AEs) were observed in 13 patients (13/20, 65%), and 1 patient had a grade 5 AE. The most frequent grade 3 AE was lymphopenia (12/13, 92%). Eighteen patients underwent surgery within 4-9 weeks after PPCT and the pCR rate was 55.6% (10/18).

This study (PALACE-2) will evaluate the efficacy of preoperative pembrolizumab with concurrent chemoradiotherapy in patients with locally advanced esophageal squamous cell carcinoma in multicentres.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in this study only if ALL of the following criteria apply:

1. Histologically confirmed cT2-T4a,N0-N+,M0 resectable esophageal squamous cell carcinoma.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
3. Patients approve and sign the informed consent

Exclusion Criteria:

1. Patients with active autoimmune disease or history of autoimmune disease.
2. Patients who have a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications.
3. Subjects with a history of symptomatic interstitial lung disease.
4. History of allergy to study drug components.
5. Women must not be pregnant or breast-feeding.
6. Men with female partners (WOCBP) that are not willing to use contraception.
7. Patient has received prior chemotherapy, radiotherapy, target therapy and immune therapy for this malignancy or for any other past malignancy.
8. Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response | 1 month after resection
  Pathologic complete response was defined as pT0N0M0

SECONDARY OUTCOMES:
3-year disease free survival | 3 years after resection
  Percentage of Participants With 3-Year disease-Free Survival (DFS), as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST)1.1. Disease free survival defined as the time from enrollment to the first documented disease progression of local recurrence or distant metastasis or death due to any cause.
Overall Survival (OS) | 5 years
  OS is defined as the time from enrollment to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Hecheng Li, MD&PHD, Principal Investigator — Ruijin hospitalRuijin Hospital, Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zheng Y, Li C, Yu B, Zhao S, Li J, Chen X, Li H. Preoperative pembrolizumab combined with chemoradiotherapy for esophageal squamous cell carcinoma: Trial design. JTCVS Open. 2021 Nov 10;9:293-299. doi: 10.1016/j.xjon.2021.11.003. eCollection 2022 Mar. PMID 36003437
- [Derived] Li C, Zhao S, Zheng Y, Han Y, Chen X, Cheng Z, Wu Y, Feng X, Qi W, Chen K, Xiang J, Li J, Lerut T, Li H. Preoperative pembrolizumab combined with chemoradiotherapy for oesophageal squamous cell carcinoma (PALACE-1). Eur J Cancer. 2021 Feb;144:232-241. doi: 10.1016/j.ejca.2020.11.039. Epub 2020 Dec 26. PMID 33373868